CLINICAL TRIAL: NCT05296447
Title: A Long-term Follow-Up Study to Evaluate the Safety and Efficacy of Suprachoroidal Administration of RGX-314 for Diabetic Retinopathy Without Center Involved-Diabetic Macular Edema
Brief Title: Long-Term Follow-Up Study of RGX-314 Administered in the Suprachoroidal Space for Participants With Diabetic Retinopathy
Status: Enrolling by invitation | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-314-5201
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy, DR
Keywords: Diabetic Retinopathy, DR
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Roll Over: No intervention - all subjects that previously received RGX-314 in a parent study
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — All subjects that previously received RGX-314 in a parent study

SUMMARY:
This is a prospective, observational study designed to evaluate the long-term safety and efficacy of RGX-314. Eligible participants are those who were previously enrolled in a clinical study of DR without center involved-diabetic macular edema (CI-DME) in which they received SCS administration of RGX-314. Enrollment of each participant in the current study should occur after the participant has completed either the end of study or early discontinuation visit in the previous (parent) clinical study. Participants will be followed for a total of 5 years post-RGX-314 administration (inclusive of the parent study). As such, the total study duration for each participant may vary depending on when they enroll in the current study following RGX-314 administration in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written, signed informed consent for this study
* Must have been enrolled in a previous clinical study of RGX-314 for the treatment of DR without CI-DME and must have received an SCS injection of RGX-314 in that study
* Must be willing and able to comply with all study procedures

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes participants who received RGX-314 in a parent study of DR without center involved-diabetic macular edema
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety of RGX-314 | 5 years inclusive of the parent study
  Incidence of overall and ocular adverse events, serious adverse events, and all adverse events of special interest

SECONDARY OUTCOMES:
Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in DR by ETDRS-DRSS on 4-widefield digital stereoscopic fundus photography | 5 years, inclusive of the parent study
Proportion of participants achieving 0-step (no change), a 1-step or greater, a 2-step or greater, or a 3-step or greater improvement in DR per ETDRS-DRSS on 4-widefield digital stereoscopic fundus photography from baseline | 5 years, inclusive to the parent study
Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in BCVA | 5 years, inclusive to the parent study
Proportion of participants gaining or losing ≥5, 10 and 15 letters in BCVA compared with baseline (ie, prior to RGX-314 administration in the parent study) | 5 years, inclusive to the parent study
Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in central subfield thickness as measured by SD-OCT | 5 years, inclusive to the parent study
Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in the area of retinal nonperfusion on ultra-widefield Optos FA | 5 years, inclusive to the parent study
Proportion of participants requiring any additional intervention for ocular diabetic complications (eg, anti-VEGF intravitreal injection or PRP) | 5 years, inclusive to the parent study
Proportion of participants with any sight-threatening ocular diabetic complications | 5 years, inclusive to the parent study

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - American Institute of Research, Los Angeles, California
  - Northern California Retina Vitreous Associates Medical Group Inc, Mountain View, California
  - California Eye Specialists Medical Group, Inc, Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - California Retina Consultants CRC, Santa Barbara, California
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Sierra eye Associates, Reno, Nevada
  - New Jersey Retina, Teaneck, New Jersey
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
  - Retinovitreous Associates, LTD, Philadelphia, Pennsylvania
  - Charles Retina Institute, P.C, Germantown, Tennessee
  - Austin Clinical Research, Austin, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No